CLINICAL TRIAL: NCT00914836
Title: Comparison of 2 Doses of Corticosteroid Subacromial Injections for the Treatment of Painful Shoulder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in the department
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: orit semana, haemek medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-09
Record Dates: First submitted 2009-05-17; First posted 2009-06-05 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Tendonitis; Bursitis
Keywords: shoulder; subacromion; corticosteroid; bursitis; tendinitis; calcific tendonitis; subacromial bursitis; rotator cuff tendinitis
MeSH Terms: conditions — Tendinopathy; Bursitis; Rotator Cuff Injuries | interventions — betamethasone sodium phosphate; betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 cc - Betamethasone Sodium Phosphate (Active Comparator): 1 cc - Betamethasone Sodium Phosphate
  Interventions: Drug: Betamethasone Sodium Phosphate; Drug: 1 cc - Betamethasone Sodium Phosphate
- 2 cc - Betamethasone Sodium Phosphate (Active Comparator): 2 cc - Betamethasone Sodium Phosphate
  Interventions: Drug: Betamethasone Sodium Phosphate; Drug: 2 cc - Betamethasone Sodium Phosphate

INTERVENTIONS:
Drug: Betamethasone Sodium Phosphate — 1cc:2cc
  Other Names: diprospan
Drug: 1 cc - Betamethasone Sodium Phosphate — Betamethasone Sodium Phosphate
  Other Names: diprospan
  Arms: 1 cc - Betamethasone Sodium Phosphate
Drug: 2 cc - Betamethasone Sodium Phosphate — Betamethasone Sodium Phosphate
  Other Names: diprospan
  Arms: 2 cc - Betamethasone Sodium Phosphate

SUMMARY:
The use of corticosteroid subacromial injections have been found to be effective for the treatment of shoulder pain. Higher doses may be better than lower doses for subacromial corticosteroid injection for rotator cuff tendonitis. The investigators aim this study to compare 2 doses of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* subacromial bursitis
* tendinitis
* Calcific Tendonitis

Exclusion Criteria:

* rotator cuff tear
* osteoarthritis
* pregnancy
* local or systemic infection
* steroid or lidocaine sensitivity

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
constant score | 9 month

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

REFERENCES:
- [Background] van der Heijden GJ, van der Windt DA, Kleijnen J, Koes BW, Bouter LM. Steroid injections for shoulder disorders: a systematic review of randomized clinical trials. Br J Gen Pract. 1996 May;46(406):309-16. PMID 8762750